CLINICAL TRIAL: NCT05605522
Title: A Phase 1 Study of [225Ac]-FPI-2059 in Adult Participants With NTSR1-Expressing Advanced, Metastatic and/or Recurrent Solid Tumours
Brief Title: A Study of [225Ac]-FPI-2059 in Adult Participants With Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor reprioritization of active trials.
Sponsor: 3B Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FPI-2059-101
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Squamous Cell Carcinoma of Head and Neck; Colorectal Cancer; Gastric Cancer; Ewing Sarcoma; NTSR1 Expressing Solid Tumours; Neuroendocrine Differentiated (NED) Prostate Cancer
Keywords: Solid Tumor; FPI-2059; FPI-2058; Pancreas; Prostate; Neuroendocrine; Stomach cancer; Gastric; Ewing sarcoma; HNSCC; Squamous cell carcinoma; CRC; Colorectal; actinium; targeted alpha therapy; radiopharmaceuticals
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Stomach Neoplasms; Sarcoma, Ewing; Prostatic Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental)
  Interventions: Drug: [225]-FPI-2059; Drug: [111In]-FPI-2058
- Phase 1 Dose Expansion (Experimental)
  Interventions: Drug: [225]-FPI-2059; Drug: [111In]-FPI-2058

INTERVENTIONS:
Drug: [225]-FPI-2059 — [225Ac]-FPI-2059 is a targeted alpha therapeutic that consists of an NTSR1-targeting small molecule that is linked to Ac-225, an alpha particle emitting radionuclide. Participants will be dosed through IV administration every 56 days up to four cycles. The dose depends on cohort assignment.
  In the Dose Expansion arm, [225Ac]-FPI-2059 will be administered at the RP2D as determined in Phase 1 Dose Escalation.
Drug: [111In]-FPI-2058 — [111In]-FPI-2058 is an imaging agent that consists of an NTSR1-targeting small molecule linked to In-111.Participants will receive [111In]-FPI-2058 by IV Injection for imaging once during screening period. The dose is consistent across cohorts.

SUMMARY:
This is a first-in-human Phase 1 clinical trial designed to investigate the safety, tolerability, pharmacokinetics, and biodistribution of [225Ac]-FPI-2059 and [111In]-FPI-2058 in participants with neurotensin receptor 1 (NTSR1)-expressing solid tumours.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, non-randomized, multi-centre, open-label clinical trial designed to investigate the safety, tolerability, dosimetry, biodistribution, and pharmacokinetics (PK) of [225Ac]-FPI-2059 and [111In]-FPI-2058, as well as the pharmacodynamics and preliminary anti-tumour activity of [225Ac]-FPI-2059 in participants with neurotensin receptor 1 (NTSR1)-expressing advanced, metastatic and/or recurrent solid tumours.

The study will employ a 3+3 dose escalation design to identify the recommended phase 2 dose (RP2D) and regimen of [225Ac]-FPI-2059 administered intravenously every 56 days.

After the RP2D for [225Ac]-FPI-2059 is determined, enrolment will continue into an expansion cohort, to confirm the safety and tolerability of the RP2D, as well as to identify any preliminary evidence of efficacy in selected NTSR1-expressing tumour types.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed ICF prior to initiation of any study-specific procedures
* Histologically and/or cytologically confirmed solid tumor that is metastatic or locally advanced, inoperable, or recurrent. Solid tumors indications may include PDAC, CRC, NED prostate cancer, gastric cancer, SCCHN, and Ewing sarcoma.
* Disease that has progressed despite prior treatment, and for which additional effective standard therapy is not available or is contraindicated, not tolerable, or the patient refuses standard therapy
* Measurable disease per RECIST v.1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Sufficient target expression in at least one measurable lesion as determined by imaging following injection of [111In]-FPI-2058
* Adequate organ function
* Tumor tissue (either archival within the last 24 months or fresh biopsy)

Key Exclusion Criteria:

* Previous treatment with any radiopharmaceutical
* Contraindications to or inability to perform the imaging procedures required in this study
* Anti-cancer therapy, such as chemotherapy, immunotherapy, hormonal therapy, targeted therapy, or investigational agents within certain amount of time prior to administration of the first dose of [111In]-FPI-2058
* Radiation therapy (RT) within 28 days prior to the first dose of [111In]-FPI-2058
* Patients with known CNS metastatic disease
* Concurrent severe and/or uncontrolled illness that would limit compliance with study requirements
* Known or suspected allergies or contraindication to the investigational treatment
* Received any type of vaccine within 30 days prior to the first dose of [111In]-FPI-2058

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events to evaluate safety and tolerability of [225Ac]-FPI-2059 and [111In]-FPI-2058 | approximately 5 years post final administration
Maximum tolerated dose (MTD) of [225Ac]-FPI-2059 | 56 days post administration
Radiation dose of [111In]-FPI-2058 and [225Ac]-FPI-2059 to whole body, organs, and selected regions of interest | within 56 days of administration

SECONDARY OUTCOMES:
Anti-tumor activity of [225Ac]-FPI-2059 regimen measured by response per RECIST v1.1 | approximately 5 years post final administration
Tumor uptake of [111In]-FPI-2058 by evaluating SPECT/CT and planar images | within 56 days of administration
Pharmacokinetics (PK) of [225Ac]-FPI-2059 and [111In]-FPI-2059 by measuring changes in clearance, AUC, Cmax, and half-life | approximately 36 days of final administration

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Enke, Study Director — 3B Pharmaceuticals GmbH
Locations (8):
- United States (7):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - City of Hope Medical Center, Duarte, California
  - Hoag Family Cancer Institute, Newport Beach, California
  - University of Kentucky, Lexington, Kentucky
  - Advanced Molecular Imaging and Therapy, Glen Burnie, Maryland
  - Washington University, St Louis, Missouri
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
- Westmead Hospital, Sydney, New South Wales, Australia